CLINICAL TRIAL: NCT04221451
Title: A Multicenter, Multinational, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy, Pharmacodynamics, Pharmacokinetics, Safety, and Tolerability of Venglustat in Late-onset GM2 Gangliosidosis (Tay-Sachs Disease and Sandhoff Disease) Together With a Separate Basket for Juvenile/Adolescent Late-onset GM2 Gangliosidosis and Ultra-rare Diseases Within the Same and Similar Glucosylceramide-based Sphingolipid Pathway
Brief Title: A Multinational, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy, Pharmacodynamics, Pharmacokinetics, and Safety of Venglustat in Late-onset GM2
Acronym: AMETHIST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Discontinued based on the absence of positive trends on clinical endpoints.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC15299; U1111-1197-7905 (Registry Identifier: ICTRP); EFC15299 (Other: Sanofi Identifier); 2019-002375-34 (EudraCT Number)
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Tay-Sachs Disease; Sandhoff Disease
MeSH Terms: conditions — Tay-Sachs Disease; Sandhoff Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GZ402671 (Experimental): Primary population: participant will receive venglustat dose once daily during the primary analysis period (104 weeks) and the open-label extension period (104 weeks).
  Secondary population: participant will receive venglustat at various doses once daily during the primary analysis period open-label (104 weeks) and the open-label extension period (104 weeks).
  Interventions: Drug: venglustat GZ402671
- Placebo (Placebo Comparator): Primary population: participants will receive placebo once daily during the primary analysis period (104 weeks) and will receive venglustat dose once daily during the open-label extension period (104 weeks).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: venglustat GZ402671 — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: GZ402671
Drug: placebo — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Placebo

SUMMARY:
Primary Objectives:

Primary population (adult participants with late-onset GM2 gangliosidosis): To assess the efficacy and pharmacodynamics (PD) of daily oral dosing of venglustat when administered over a 104-week period

Secondary population (participants with juvenile/adolescent late-onset GM2 gangliosidosis, GM1 gangliosidosis, saposin C deficiency, sialidosis type 1 or juvenile/adult galactosialidosis): To assess PD response (plasma and CSF GL-1 biomarker and disease specific biomarkers) of venglustat when administered once daily over a 104-week period

Secondary Objectives:

Primary population:

* To assess the PD of daily oral dosing of venglustat and the effect of venglustat on selected performance test and scale over a 104-week period
* To determine the safety and tolerability of venglustat when administered orally once daily over a 104-week period
* To assess the pharmacokinetics (PK) of venglustat in plasma and cerebrospinal fluid (CSF)

Secondary population:

* To assess the effect of venglustat on selected performance tests and scale over a 104-week period
* To determine the safety and tolerability of venglustat when administered once daily over a 104-week period
* To assess the PK of venglustat in plasma and CSF
* To assess the acceptability and palatability of the venglustat tablet

DETAILED DESCRIPTION:
The total duration is up to approximately 223 weeks, including a 60-day screening period, a 104-week primary analysis treatment period, a 104-week open-label extension treatment period and a 6-week post-treatment safety observation period.

ELIGIBILITY:
Inclusion criteria :

* Primary population and adult secondary population: age ≥ 18 years
* Juvenile/adolescent secondary population: 2 ≥ age < 18 years with weight ≥ 10 kg
* Participants with a diagnosis of late onset GM2 gangliosidosis (Tay-Sachs disease and Sandhoff disease) caused by genetic β-hexosaminidase deficiency resulting from mutations in the HEXA or HEXB genes (primary population only); a secondary population will enroll patients with diagnosis of juvenile/adolescent GM2 gangliosidosis, GM1 gangliosidosis, saposin C deficiency, sialidosis type 1 or juvenile adult galactosialidosis
* For primary population, the participant has the ability to perform the 9-HPT at the screening visit in < = 240 seconds for the 2 consecutive trials of the dominant hand and the 2 consecutive trials of the nondominant hand.
* Participants with a history of seizures well controlled by medication other than strong or moderate inducer or inhibitor of CYP3A4
* Participant is cooperative, able to ingest oral medication, willing to travel to a study site (if applicable), and able to comply with all aspects of the study, including all assessments, according to the Investigator's judgement
* Signed written informed assent/consent
* Contraception for sexually active male participants or female patient; not pregnant or breastfeeding; no sperm donating for male participant

Exclusion criteria:

* Participant has clinical features of Tay-Sachs or Sandhoff disease, not caused by β-hexosaminidase deficiency resulting from mutations in the HEXA or HEXB genes and/or is without clinical features
* For primary population and participants with juvenile/adolescent late onset GM2 gangliosidosis and GM1 gangliosidosis, the participant cannot understand and perform all age-appropriate study assessments with the exception of 25FWT and PROs.
* Relevant medical disorders that would compromise his/her safety
* Documented diagnosis of hepatitis B, C, human immunodeficiency virus 1 or 2
* World Health Organization (WHO) grade >= 2 cortical cataract or a grade >= 2 posterior subcapsular cataract; patients with nuclear cataracts will be accepted
* Participant who requires invasive ventilatory support
* Current treatment by anticoagulants, cataractogenic medications or any medications that may worsen the vision of patient with cataract
* Previous treatment with substrate reduction therapy (SRT) within 3 months prior to study enrollment, strong or moderate inducers or inhibitors of CYP3A4 within 14 days or 5 half-lives prior to enrollment. This also includes the consumption of grapefruit, grapefruit juice or grapefruit products within 72hrs prior to starting investigational medicinal product (IMP) administration.
* Current participation in another study
* Use of investigational medicinal product (IMP) within 3 months or 5 half-lives, whichever is longer, before study enrollment (for N-acetyl-leucine, within 5 half-lives before study enrollment).
* Liver enzymes (alanine aminotransferase [ALT]/aspartate aminotransferase [AST]) or total bilirubin > 2 x the upper limite of normal (ULN) at the time of screening unless the participant has the diagnosis of Gilbert syndrome and maintains a level of bilirubin < 5 mg/dl and direct bilirubin < 20% (1 mg/dl) of total bilirubin level
* Renal insufficiency is defined by estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2 at the screening visit

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2024-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (23):
- United States (5):
  - Ataxia Center and HD Center of Excellence, 300 UCLA Med Plaza, Suite B200 - Investigational site number 8400004, Los Angeles, California
  - Emory Genetics - Investigational site number 8400006, Atlanta, Georgia
  - NIH National Human Genome Research Institute - 10 Center Dr - Bldg. 10 CRC3-2551 MSC 1205 - Investigational site number 8400005, Bethesda, Maryland
  - Massachusetts General Hospital - Charles River Plaza 175 Cambridge St. Ste 340 - Investigational site number 8400002, Boston, Massachusetts
  - NYU Langone - 550 First Avenue-Investigational site number 8400001, New York, New York
- Argentina (2):
  - Hospital Universitario Austral Pilar, Buenos Aires_Unidad de Investigación Clínica_investigational site number 0320002, Pilar, Buenos Aires
  - Clínica Universitaria Reina Fabiola Córdoba_investigational site number 0320001, Córdoba
- Hospital de Clinicas de Porto Alegre _investigational site number 0760001, Porto Alegre, Rio Grande do Sul, Brazil
- Vseobecna Fakultni Nemocnice V Praze Metabolicke centrum U Nemocnice 2_investigational site number 2030001, Prague, Czechia
- APHP - Centre Hospitalier la Pitié Salpetrière, Service de Neurologie, 47-83 Boulevard De l'Hôpital_Investigational site number 2500001, Paris, France
- Universitätsklinikum der Justus-Liebig-Universität Gießen Zentrum für Kinderheilkunde und Jugendmedizin Feulgenstraße 10-12_investigational site number 2760001, Giessen, Germany
- Investigational Site Number : 3800001, Milan, Italy
- Japan (2):
  - Japanese Red Cross Akita Hospital 222-1 Nawashirosawa, Kamikitatesaruta_investigational site number 3920001, Akita, Akita
  - Tohoku Medical and Pharmaceutical University Hospital_investigation site number 3920002, Sendai, Miyagi
- Centro Hospitalar Universitário Lisboa Norte- Hospital Santa Maria Avenida Professor Egas Moniz_investigational site number 6200002, Lisbon, Portugal
- Research Center Of Neurology 80, Volokolamskoye shosse_investigational site number 6430001, Moscow, Russia
- Spain (3):
  - Hospital Universitari de Bellvitge. Feixa Llarga, S / N_investigational site number 7240004, L'Hospitalet de Llobregat, Barcelona [Barcelona]
  - Hospital Maternoinfantil Sant Joan de Déu Paseo de Sant Joan de Déu, 2_investigational site number 7240001, Esplugues de Llobregat, Catalunya [Cataluña]
  - Hospital Clínico Universitario de Santiago-CHUS. Travesia de Chopuana, s/n_investigational site number 7240002, Santiago de Compostela, Galicia [Galicia]
- Gazi Universitesi Tip Fakultesi Emniyet Street Mevlana Blv Besevler Yenimahalle_investigational site number 7920001, Ankara, Turkey (Türkiye)
- United Kingdom (3):
  - Cambridge University Hospitals NHS Foundation Trust Addenbrookes Hospital Hills Road_investigational site number 8260001, Cambridge, Cambridgeshire
  - Investigational Site Number : 8260003, Manchester
  - Salford Royal NHS Foundation Trust Salford Royal Hospital Stott Lane_investigational site number 8260002, Salford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Nicoli ER, Annunziata I, d'Azzo A, Platt FM, Tifft CJ, Stepien KM. GM1 Gangliosidosis-A Mini-Review. Front Genet. 2021 Sep 3;12:734878. doi: 10.3389/fgene.2021.734878. eCollection 2021. PMID 34539759
- See also: EFC15299 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25230&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 2 periods: primary analysis period (PAP) & open-label extension (OLE) period. In PAP, primary population (PP) was randomized in a 2:1 ratio to receive either venglustat or placebo in double-blind manner. Secondary population (SP) received OL venglustat. Post completion of PAP, eligible participants entered OLE in which all participants received OL venglustat. The study was early terminated based on absence of positive trends on clinical endpoints; no safety concerns.
Pre-assignment Details: In PAP, 59 participants in the PP (adult participants with diagnosis of late-onset disialotetrahexosylganglioside [GM2] gangliosidosis) and 16 participants in the SP (juvenile/adolescent participants with diagnosis of late-onset GM2 gangliosidosis, monosialotetrahexosylganglioside [GM1] gangliosidosis, saposin C deficiency, sialidosis type 1, or juvenile/adult galactosialidosis) were treated. Randomization for PP was stratified on participant's ability to walk at baseline visit (yes/no).
Groups:
- PAP: PP: Placebo: Participants in PP received placebo matched to venglustat oral tablet once daily for 104 weeks in a double-blind manner in PAP.
- PAP: PP: Venglustat: Participants in PP received venglustat 15 milligrams (mg) oral tablet once daily for 104 weeks in a double-blind manner in PAP.
- PAP: SP: Venglustat: Participants in SP received venglustat oral tablet once daily based on the body weight for 104 weeks in an open-label manner in PAP as follows:
  15 mg if >=50 kilograms [kg], 12 mg if 30 kg to <50 kg, 6 mg if 15 kg to <30 kg and 4 mg if 10 kg to <15 kg.
- OLE: PP: Delayed Venglustat: Participants in PP who previously received placebo in PAP received venglustat 15 mg oral tablet once daily for 104 weeks in an open-label manner in OLE.
- OLE: PP: Early Venglustat: Participants in PP who previously received venglustat in PAP continued to receive venglustat 15 mg oral tablet once daily for 104 weeks in an open-label manner in OLE.
- OLE: SP: Venglustat: Participants in SP who previously received venglustat in PAP continued to receive venglustat oral tablet once daily based on the body weight for 104 weeks in an open-label manner in OLE as follows:
  15 mg if >=50 kg, 12 mg if 30 kg to <50 kg, 6 mg if 15 kg to <30 kg and 4 mg if 10 kg to <15 kg.
Period: PAP: Baseline (Day 1) up to 104 Weeks
Arm/Group | PAP: PP: Placebo | PAP: PP: Venglustat | PAP: SP: Venglustat | OLE: PP: Delayed Venglustat | OLE: PP: Early Venglustat | OLE: SP: Venglustat
Started | 19 | 40 | 16 | 0 | 0 | 0
Completed (PAP period) | 17 | 35 | 14 | 0 | 0 | 0
Not Completed | 2 | 5 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0
Period: OLE (104 Weeks): From 104 to 208 Weeks
Arm/Group | PAP: PP: Placebo | PAP: PP: Venglustat | PAP: SP: Venglustat | OLE: PP: Delayed Venglustat | OLE: PP: Early Venglustat | OLE: SP: Venglustat
Started (Only eligible participants entered the OLE period) | 0 | 0 | 0 | 16 | 34 | 14
Completed (OLE period) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 16 | 34 | 14
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 1 | 2
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 13 | 33 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population included all participants from screened population who were allocated to a randomized study drug by interactive response technology regardless of whether the study drug was received or not.
Groups:
- PAP: PP: Venglustat: Participants in PP received venglustat 15 mg oral tablet once daily for 104 weeks in a double-blind manner in PAP.
- PAP: SP: Venglustat: Participants in SP received venglustat oral tablet once daily based on the body weight for 104 weeks in an open-label manner in PAP as follows:
  15 mg if >=50 kg, 12 mg if 30 kg to <50 kg, 6 mg if 15 kg to <30 kg and 4 mg if 10 kg to <15 kg.
- Total: Total of all reporting groups
Arm/Group | PAP: PP: Placebo | PAP: PP: Venglustat | PAP: SP: Venglustat | Total
Number analyzed (Participants) | 19 | 40 | 16 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (15.4) | 37.0 (13.3) | 12.4 (7.3) | 32.0 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 19 | 11 | 40
  Male | 9 | 21 | 5 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 17 | 35 | 12 | 64
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 5
PP: Cerebrospinal fluid (CSF) GM2 biomarker [Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)] — Lumbar puncture was performed for obtaining CSF samples at baseline to assess the presence of GM2 biomarker in PP in PAP. Population: PAP: Primary pharmacodynamic (PD) population included all randomized participants with diagnosis of late-onset GM2 gangliosidosis aged >=18 years who received at least 1 dose of study drug and who had baseline and post-baseline assessments of PD. Only those PP participants with data collected at baseline are reported.
  nanogram/milliliter (ng/mL)
    number analyzed (Participants) | 18 | 39 | 0 | 57
    (all) | 67.11 (34.15) | 63.00 (36.84) |  | 64.30 (35.76)
PP: 9-hole peg Test (9-HPT) [Mean (Standard Deviation); unit: seconds] — 9-HPT is a test of upper extremity (arm and hand) function.Participant is seated at table with small, shallow container holding pegs & block containing 9 empty holes.When stopwatch is started,participant picks up 9 pegs one at a time as quickly as possible,puts them in 9 holes and removes them again as quickly as possible one at a time,replacing them into shallow container; 2 trials for each hand. Total time (ranging up to 300 seconds):averaged, converted to reciprocals which were averaged and back-transformed to obtain global 9-HPT.Higher value on 9-HPT is indicative of higher disability. Population: Only PP participants are included for this analysis.
  seconds
    number analyzed (Participants) | 19 | 40 | 0 | 59
    (all) | 45.89 (34.65) | 41.93 (26.56) |  | 43.20 (29.16)
Clinical diagnosis of SP [Count of Participants; unit: Participants] — Participants with clinical diagnosis of juvenile/adolescent GM2 gangliosidosis, monosialotetrahexosylganglioside (GM1) gangliosidosis, sialidosis type 1, juvenile/adult galactosialidosis, or saposin C deficiency were referred to as SP. Population: Only SP participants are included for this analysis.
  Participants
    number analyzed (Participants) | 0 | 0 | 16 | 16
    Juvenile/adolescent GM2 gangliosidosis |  |  | 7 | 7
    GM1 gangliosidosis |  |  | 7 | 7
    Saposin C deficiency |  |  | 0 | 0
    Sialidosis type 1 |  |  | 1 | 1
    Juvenile/adult galactosialidosis |  |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: PAP: PP: Percent Change From Baseline in CSF GM2 Biomarker to Week 104
Description: Lumbar puncture was performed for obtaining CSF samples at specified timepoints to assess the presence of GM2 biomarker in PP in PAP. The baseline value was defined as the last available value before or equal to the first dose of study drug date in the PAP.
Time Frame: Baseline (Day 1) and Week 104
Population: PAP: Primary PD population included all randomized participants with diagnosis of late-onset GM2 gangliosidosis aged >=18 years who received at least 1 dose of study drug and who had baseline and post-baseline assessments of PD. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | PAP: PP: Placebo | PAP: PP: Venglustat
Number analyzed (Participants) | 16 | 31
percent change | -11.33 (4.23) | -47.57 (3.04)
Statistical Analysis 1: Comparison: PAP: PP: Placebo vs PAP: PP: Venglustat; Mean percent change from baseline obtained from robust analysis of covariance (ANCOVA) using Huber's M estimation, including the fixed categorical effects of treatment (venglustat versus placebo) and the continuous fixed covariate of baseline value; Test type: Superiority; p < 0.0001, Robust ANCOVA; Mean difference = -36.24, 90% CI 2-sided [-44.80 to -27.68], Standard Error of Mean 5.20

2. Primary Outcome: PAP: PP: Annualized Rate of Change From Baseline in the 9-HPT to Week 104
Description: 9-HPT is a test of upper extremity (arm and hand) function.Participant is seated at table with small, shallow container holding pegs and block containing 9 empty holes.On start command when stopwatch is started,participant picks up 9 pegs one at a time as quickly as possible, puts them in 9 holes and once they are in holes, removes them again as quickly as possible one at a time,replacing them into shallow container. Both dominant and non-dominant hands are tested twice (2 consecutive trials of dominant hand followed immediately by 2 consecutive trials of non-dominant hand).Total time (ranging up to 300 seconds):averaged, converted to reciprocals which were averaged and back-transformed to obtain global 9-HPT.Higher value on 9-HPT is indicative of higher disability.Mean annualized rate of change in 9-HPT was obtained from exponential transformation of mean slope of log-transformed 9-HPT.Baseline: last available value before or equal to the first dose of study drug date in the PAP.
Time Frame: Baseline (Day 1) and Week 104
Population: PAP: Primary efficacy population included all randomized participants with diagnosis of late-onset GM2 gangliosidosis aged >=18 years. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Error); unit: percent per year
Arm/Group | PAP: PP: Placebo | PAP: PP: Venglustat
Number analyzed (Participants) | 18 | 39
percent per year | 0.95 (1.92) | 2.49 (1.35)
Statistical Analysis 1: Comparison: PAP: PP: Placebo vs PAP: PP: Venglustat; Mean slope of log-transformed 9-HPT obtained from a robust ANCOVA on individual slopes of log-transformed 9-HPT using Huber's M estimation; Test type: Superiority; p = 0.7435, Robust ANCOVA; The robust ANCOVA included fixed effect of treatment (venglustat versus placebo) and continuous fixed covariate of log-transformed baseline value; Mean difference = 1.54, 90% CI 2-sided [-2.33 to 5.39], Standard Error of Mean 2.35

3. Primary Outcome: PAP: SP: Percent Change From Baseline in Plasma and CSF Biomarkers (Glucosylceramide [GL-1] and GM2) to Week 104 in Juvenile/Adolescent Late-onset GM2 Gangliosidosis Participants
Description: Plasma and CSF samples were collected at specified timepoints to assess the presence of GL-1 and GM2 biomarkers in juvenile/adolescent late-onset GM2 gangliosidosis participants of SP in PAP. The baseline value was defined as the last available value before or equal to the first dose of study drug date in the PAP.
Time Frame: Baseline (Day 1) and Week 104
Population: PAP: Analysis was performed on juvenile/adolescent late-onset GM2 gangliosidosis participants from secondary PD population which included all enrolled participants with this clinical diagnosis who received at least 1 dose of study drug and who had baseline and post-baseline assessments of PD.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PAP: SP: Venglustat
Number analyzed (Participants) | 7
percent change
  GL-1: CSF | -82.35 (9.94)
  GL-1: Plasma | -79.28 (2.56)
  GM2: CSF | -43.41 (23.14)
  GM2: Plasma | -55.91 (11.76)

4. Primary Outcome: PAP: SP: Percent Change From Baseline in Plasma and CSF GL-1 and GM1 Biomarkers to Week 104 in GM1 Gangliosidosis Participants
Description: Plasma and CSF samples were collected at specified timepoints to assess the presence of GL-1 and GM1 biomarkers in GM1 gangliosidosis participants of SP in PAP. The baseline value was defined as the last available value before or equal to the first dose of study drug date in the PAP.
Time Frame: Baseline (Day 1) and Week 104
Population: PAP: Analysis was performed on GM1 gangliosidosis participants from secondary PD population which included all enrolled participants with this clinical diagnosis who received at least 1 dose of study drug and who had baseline and post-baseline assessments of PD. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PAP: SP: Venglustat
Number analyzed (Participants) | 6
percent change
  GL-1: CSF: number analyzed (Participants) | 4
  GL-1: CSF | 17.42 (188.41)
  GL-1: Plasma | -80.42 (8.17)
  GM1: CSF: number analyzed (Participants) | 4
  GM1: CSF | -32.35 (17.46)
  GM1: Plasma | -52.32 (16.76)

5. Primary Outcome: PAP: SP: Percent Change From Baseline in Plasma and CSF GL-1, GM2 and Monosialodihexosylganglioside (GM3) Biomarkers to Week 104 in Sialidosis Type 1 Participant
Description: Plasma and CSF samples were collected at specified timepoints to assess the presence of GL-1, GM2 and GM3 biomarkers in sialidosis type 1 participant of SP in PAP. The baseline value was defined as the last available value before or equal to the first dose of study drug date in the PAP. Analysis was planned to be performed on sialidosis type 1 participant from secondary PD population (all enrolled participants with this clinical diagnosis who received at least 1 dose of study drug and who had baseline and post-baseline assessments of PD).
Time Frame: Baseline (Day 1) and Week 104
Population: Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with sialidosis type 1 was enrolled in the study.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PAP: SP: Venglustat
Number analyzed (Participants) | 1
percent change
  GL-1: CSF | NA — Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with sialidosis type 1 was enrolled in the study.
  GL-1: Plasma | NA — Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with sialidosis type 1 was enrolled in the study.
  GM2: CSF | NA — Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with sialidosis type 1 was enrolled in the study.
  GM2: Plasma | NA — Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with sialidosis type 1 was enrolled in the study.
  GM3: CSF | NA — Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with sialidosis type 1 was enrolled in the study.
  GM3: Plasma | NA — Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with sialidosis type 1 was enrolled in the study.

6. Primary Outcome: PAP: SP: Percent Change From Baseline in Plasma and CSF GL-1, GM1 and GM3 Biomarkers to Week 104 in Juvenile/Adult Galactosialidosis Participants
Description: Plasma and CSF samples were collected at specified timepoints to assess the presence of GL-1, GM1 and GM3 biomarkers in juvenile/adult galactosialidosis participants of SP in PAP. The baseline value was defined as the last available value before or equal to the first dose of study drug date in the PAP. Analysis was planned to be performed on juvenile/adult galactosialidosis participant from secondary PD population which included all enrolled participants with this clinical diagnosis who received at least 1 dose of study drug and who had baseline and post-baseline assessments of PD.
Time Frame: Baseline (Day 1) and Week 104
Population: Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with juvenile/adult galactosialidosis was enrolled in the study.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PAP: SP: Venglustat
Number analyzed (Participants) | 1
percent change
  GL-1: CSF | NA — Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with juvenile/adult galactosialidosis was enrolled in the study.
  GL-1: Plasma | NA — Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with juvenile/adult galactosialidosis was enrolled in the study.
  GM1: CSF | NA — Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with juvenile/adult galactosialidosis was enrolled in the study.
  GM1: Plasma | NA — Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with juvenile/adult galactosialidosis was enrolled in the study.
  GM3: CSF | NA — Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with juvenile/adult galactosialidosis was enrolled in the study.
  GM3: Plasma | NA — Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with juvenile/adult galactosialidosis was enrolled in the study.

7. Primary Outcome: PAP: SP: Percent Change From Baseline in Plasma and CSF GL-1 Biomarker to Week 104 in Saposin C Deficiency Participants
Description: Plasma and CSF samples were planned to be collected at specified timepoints to assess the presence of GL-1 biomarkers in saposin C deficiency participants of SP in PAP. The baseline value was defined as the last available value before or equal to the first dose of study drug date in the PAP.
Time Frame: Baseline (Day 1) to Week 104
Population: PAP: Analysis was planned to be performed on saposin C deficiency participants from secondary PD population which included all enrolled participants with this clinical diagnosis who received at least 1 dose of study drug and who had baseline and post-baseline assessments of PD. As presented in baseline characteristics, there was no participant enrolled with Saposin C deficiency.
Arm/Group | PAP: SP: Venglustat
Number analyzed (Participants) | 0

8. Secondary Outcome: PAP: PP: Absolute Change From Baseline in CSF GM2 Biomarker to Week 104
Description: as for outcome 1
Time Frame: Baseline (Day 1) and Week 104
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | PAP: PP: Placebo | PAP: PP: Venglustat
Number analyzed (Participants) | 16 | 31
ng/mL | -17.64 (2.36) | -32.83 (1.70)

9. Secondary Outcome: PAP: PP and SP: Change From Baseline in 25-foot Walk Test (25FWT) to Week 104
Description: The 25FWT is a quantitative mobility and leg function performance test based on a timed 25-foot walk. The participant is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly and safely as possible for 2 trials (can use assistive devices). The time is calculated from the initiation of the instruction to start and ends when the participant has reached the 25-foot mark. The amount of time (in seconds) to walk 25 feet is recorded (ranging up to 180 seconds). The 25FWT score is defined as the average of 2 trials. A higher value on the 25FWT is indicative of higher disability. The baseline value was defined as the last available value before or equal to the first dose of study drug date in the PAP.
Time Frame: Baseline (Day 1) and Week 104
Population: PAP PP:primary efficacy population included all randomized participants with diagnosis of late-onset GM2 gangliosidosis aged >=18 years.PAP SP: secondary efficacy population included all enrolled participants with a clinical diagnosis of juvenile/adolescent late-onset GM2 gangliosidosis, GM1 gangliosidosis, saposin C deficiency, sialidosis type 1, or juvenile/adult galactosialidosis.Only those participants with ability to walk at baseline and data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | PAP: PP: Placebo | PAP: PP: Venglustat | PAP: SP: Venglustat
Number analyzed (Participants) | 16 | 30 | 11
seconds
  PP: number analyzed (Participants) | 16 | 30 | 0
  PP | 1.4 (4.2) | 8.9 (31.0) |
  SP: juvenile/adolescent late-onset GM2 gangliodosis: number analyzed (Participants) | 0 | 0 | 5
  SP: juvenile/adolescent late-onset GM2 gangliodosis |  |  | 29.6 (66.5)
  SP: GM1 gangliosidosis: number analyzed (Participants) | 0 | 0 | 6
  SP: GM1 gangliosidosis |  |  | 0.4 (0.8)
  SP: sialidosis type 1: number analyzed (Participants) | 0 | 0 | 0
  SP: juvenile/adult galactosialidosis: number analyzed (Participants) | 0 | 0 | 0
  SP: saposin C deficiency: number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: PAP: PP and SP: Change From Baseline in the Neurological Examination of the Friedreich's Ataxia Rating Scale (FARS) (FARS-neuro) to Week 104
Description: The FARS-neuro includes 23 items and is composed of 4 sections that assesses different neurological faculties: bulbar activity (4 items), upper limb coordination (5 items assessed right and left side), lower limb coordination (2 items assessed right and left side), peripheral nervous system (5 items assessed right and left side) and upright stability (7 items). Total score is calculated as the sum of scores on items of this section and ranges from 0 to 117; mean is presented. Higher value indicates higher disability. Baseline=last available value before or equal to first dose of study drug date in PAP. PP: primary efficacy population: all randomized participants with diagnosis of late-onset GM2 gangliosidosis aged >=18 years. SP: secondary efficacy population: all enrolled participants with diagnosis of juvenile/adolescent late-onset GM2 gangliosidosis, GM1 gangliosidosis, saposin C deficiency, sialidosis type 1, or juvenile/adult galactosialidosis.
Time Frame: Baseline (Day 1) and Week 104
Population: Only those participants with data collected at specified timepoints are reported. For sialidosis type 1: due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality. As presented in baseline characteristics, only 1 participant with sialidosis type 1 was enrolled in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PAP: PP: Placebo | PAP: PP: Venglustat | PAP: SP: Venglustat
Number analyzed (Participants) | 17 | 35 | 13
score on a scale
  PP: number analyzed (Participants) | 17 | 35 | 0
  PP | 0.4 (6.0) | -1.0 (8.5) |
  SP: juvenile/adolescent late-onset GM2 gangliodosis: number analyzed (Participants) | 0 | 0 | 6
  SP: juvenile/adolescent late-onset GM2 gangliodosis |  |  | 2.8 (10.6)
  SP: GM1 gangliosidosis: number analyzed (Participants) | 0 | 0 | 6
  SP: GM1 gangliosidosis |  |  | -2.5 (17.0)
  SP: sialidosis type 1: number analyzed (Participants) | 0 | 0 | 1
  SP: sialidosis type 1 |  |  | NA — Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality.
  SP: juvenile/adult galactosialidosis: number analyzed (Participants) | 0 | 0 | 0
  SP: saposin C deficiency: number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: PAP: PP and SP: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. SAE was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. TEAE were AEs that developed, worsened or became serious during the TE period.
Time Frame: From first dose of study drug (Day 1) up to end of PAP, 104 weeks
Population: PAP PP: primary safety population included all randomized participants with diagnosis of late-onset GM2 gangliosidosis aged >=18 years who received at least 1 dose of study drug.
  PAP SP: secondary safety population included all enrolled participants with a clinical diagnosis of juvenile/adolescent late-onset GM2 gangliosidosis, GM1 gangliosidosis, saposin C deficiency, sialidosis type 1, or juvenile/adult galactosialidosis, who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PAP: PP: Placebo | PAP: PP: Venglustat | PAP: SP: Venglustat
Number analyzed (Participants) | 19 | 40 | 16
Participants
  TEAEs | 19 | 40 | 14
  TESAEs | 4 | 8 | 6

12. Secondary Outcome: PAP: PP: Plasma Venglustat Concentration
Description: Plasma samples were collected at specified timepoints to obtain venglustat concentrations for PP in PAP.
Time Frame: Pre-dose (0 hour) and 0.5, 3, 8, 12 and 24 hours post-dose at Week 12
Population: PAP: Primary pharmacokinetic (PK) population included all randomized participants with diagnosis of late-onset GM2 gangliosidosis aged >=18 years who received at least 1 dose of study drug and had at least 1 PK assessment. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PAP: PP: Venglustat
Number analyzed (Participants) | 30
ng/mL
  0 hour: number analyzed (Participants) | 28
  0 hour | 112 (43.7)
  0.5 hours: number analyzed (Participants) | 27
  0.5 hours | 125 (54.1)
  3 hours | 188 (60.8)
  8 hours: number analyzed (Participants) | 29
  8 hours | 149 (47.3)
  12 hours: number analyzed (Participants) | 28
  12 hours | 132 (44.5)
  24 hours: number analyzed (Participants) | 22
  24 hours | 105 (38.5)

13. Secondary Outcome: PAP: SP: Plasma Venglustat Concentration
Description: Plasma samples were collected at specified timepoints to obtain venglustat concentration for SP in PAP. Data is presented by dose level for all diseases combined for SP in PAP.
Time Frame: Pre-dose (0 hour) and 0.5, 3, 8, 12 and 24 hours post-dose at Week 12
Population: PAP: Secondary PK population included all enrolled participants with a clinical diagnosis of juvenile/adolescent late-onset GM2 gangliosidosis, GM1 gangliosidosis, saposin C deficiency, sialidosis type 1, or juvenile/adult galactosialidosis, who received at least 1 dose of study drug and had at least 1 PK assessment. 'Overall Number of Participants Analyzed' indicates the total of maximum number of participants ('number analyzed') for each dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PAP: SP: Venglustat
Number analyzed (Participants) | 15
ng/mL
  4 mg: 0 hour: number analyzed (Participants) | 1
  4 mg: 0 hour | 56.4
  4 mg: 0.5 hours: number analyzed (Participants) | 0
  4 mg: 3 hours: number analyzed (Participants) | 1
  4 mg: 3 hours | 144
  4 mg: 8 hours: number analyzed (Participants) | 1
  4 mg: 8 hours | 101
  4 mg: 12 hours: number analyzed (Participants) | 1
  4 mg: 12 hours | 92.3
  4 mg: 24 hours: number analyzed (Participants) | 1
  4 mg: 24 hours | 58.1
  6 mg: 0 hour: number analyzed (Participants) | 7
  6 mg: 0 hour | 61.5 (34.1)
  6 mg: 0.5 hours: number analyzed (Participants) | 6
  6 mg: 0.5 hours | 85.9 (56.8)
  6 mg: 3 hours: number analyzed (Participants) | 7
  6 mg: 3 hours | 127 (72.4)
  6 mg: 8 hours: number analyzed (Participants) | 7
  6 mg: 8 hours | 97.9 (55.6)
  6 mg: 12 hours: number analyzed (Participants) | 7
  6 mg: 12 hours | 87.9 (55.9)
  6 mg: 24 hours: number analyzed (Participants) | 5
  6 mg: 24 hours | 50.2 (25.5)
  12 mg: 0 hour: number analyzed (Participants) | 4
  12 mg: 0 hour | 58.4 (40.8)
  12 mg: 0.5 hours: number analyzed (Participants) | 4
  12 mg: 0.5 hours | 67.4 (36.4)
  12 mg: 3 hours: number analyzed (Participants) | 4
  12 mg: 3 hours | 112 (40.8)
  12 mg: 8 hours: number analyzed (Participants) | 4
  12 mg: 8 hours | 98.2 (22.0)
  12 mg: 12 hours: number analyzed (Participants) | 4
  12 mg: 12 hours | 79.3 (35.8)
  12 mg: 24 hours: number analyzed (Participants) | 3
  12 mg: 24 hours | 49.5 (17.4)
  15 mg: 0 hour: number analyzed (Participants) | 3
  15 mg: 0 hour | 67.7 (7.05)
  15 mg: 1.5 hours: number analyzed (Participants) | 3
  15 mg: 1.5 hours | 86.7 (35.0)
  15 mg: 3 hours: number analyzed (Participants) | 3
  15 mg: 3 hours | 124 (16.0)
  15 mg: 8 hours: number analyzed (Participants) | 3
  15 mg: 8 hours | 96.4 (10.2)
  15 mg: 12 hours: number analyzed (Participants) | 3
  15 mg: 12 hours | 88.9 (6.05)
  15 mg: 24 hours: number analyzed (Participants) | 3
  15 mg: 24 hours | 64.5 (13.5)

14. Secondary Outcome: PAP: PP and SP: CSF Venglustat Concentration
Description: CSF samples were collected via lumbar puncture at Week 104 to obtain venglustat concentrations for PP and SP in PAP. For SP: data is presented by dose level for all diseases combined. Only those participants with data collected at specified timepoints are reported.
Time Frame: Week 104
Population: PAP: Participants (PP: primary PK population=all randomized participants with diagnosis of late-onset GM2 gangliosidosis aged >=18 years and SP: secondary PK population=all enrolled participants with diagnosis of juvenile/adolescent late-onset GM2 gangliosidosis, GM1 gangliosidosis, saposin C deficiency, sialidosis type 1, or juvenile/adult galactosialidosis) who received at least 1 dose of study drug & had at least 1 PK assessment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PAP: PP: Venglustat | PAP: SP: Venglustat
Number analyzed (Participants) | 18 | 7
ng/mL
  PP: number analyzed (Participants) | 18 | 0
  PP | 5.64 (2.05) |
  SP: 4 mg: number analyzed (Participants) | 0 | 0
  SP: 6 mg: number analyzed (Participants) | 0 | 2
  SP: 6 mg |  | 3.37 (2.19)
  SP: 12 mg: number analyzed (Participants) | 0 | 2
  SP: 12 mg |  | 3.22 (1.01)
  SP: 15 mg: number analyzed (Participants) | 0 | 3
  SP: 15 mg |  | 5.41 (0.57)

15. Secondary Outcome: PAP: PP and SP: Maximum Plasma Concentration Observed (Cmax) of Venglustat
Description: Plasma samples were collected at specified timepoints to obtain Cmax of venglustat. The mean of Cmax, irrespective of the timepoint where the patient-individual Cmax value was observed is presented as opposed to endpoint 13 wherein mean of plasma venglustat concentration at each specified timepoint is presented. For SP: data is presented by dose level for all diseases combined. Only those participants with data collected at specified timepoints are reported.
Time Frame: Pre-dose (0 hour) and 0.5, 3, 8, 12 and 24 hours post-dose at Week 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PAP: PP: Venglustat | PAP: SP: Venglustat
Number analyzed (Participants) | 30 | 15
ng/mL
  PP: number analyzed (Participants) | 30 | 0
  PP | 188 (60.8) |
  SP: 4 mg: number analyzed (Participants) | 0 | 1
  SP: 4 mg |  | 144
  SP: 6 mg: number analyzed (Participants) | 0 | 7
  SP: 6 mg |  | 127 (72.4)
  SP: 12 mg: number analyzed (Participants) | 0 | 4
  SP: 12 mg |  | 121 (39.5)
  SP: 15 mg: number analyzed (Participants) | 0 | 3
  SP: 15 mg |  | 124 (16.0)

16. Secondary Outcome: PAP: PP and SP: Time to Reach Maximum Plasma Concentration (Tmax) of Venglustat
Description: Plasma samples were collected at specified timepoints to obtain tmax of venglustat. For SP: data is presented by dose level for all diseases combined. Only those participants with data collected at specified timepoints are reported.
Time Frame: Pre-dose (0 hour) and 0.5, 3, 8, 12 and 24 hours post-dose at Week 12
Population: as for outcome 14
Measure: Median (Full Range); unit: hour
Arm/Group | PAP: PP: Venglustat | PAP: SP: Venglustat
Number analyzed (Participants) | 30 | 15
hour
  PP: number analyzed (Participants) | 30 | 0
  PP | 3.00 [2.77 to 7.05] |
  SP: 4 mg: number analyzed (Participants) | 0 | 1
  SP: 4 mg |  | 3.50
  SP: 6 mg: number analyzed (Participants) | 0 | 7
  SP: 6 mg |  | 3.00 [2.25 to 3.02]
  SP: 12 mg: number analyzed (Participants) | 0 | 4
  SP: 12 mg |  | 5.50 [3.00 to 12.00]
  SP: 15 mg: number analyzed (Participants) | 0 | 3
  SP: 15 mg |  | 3.00 [3.00 to 3.00]

17. Secondary Outcome: PAP: PP and SP: Area Under the Plasma Concentration Versus Time Curve Calculated Over a Predefined Time Period 0 to 24 Hours (AUC0-24) of Venglustat
Description: Plasma samples were collected at specified timepoints to obtain AUC0-24 of venglustat. For SP: data is presented by dose level for all diseases combined. Only those participants with data collected at specified timepoints are reported.
Time Frame: Pre-dose (0 hour) and 0.5, 3, 8, 12 and 24 hours post-dose at Week 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | PAP: PP: Venglustat | PAP: SP: Venglustat
Number analyzed (Participants) | 22 | 12
hour*ng/mL
  PP: number analyzed (Participants) | 22 | 0
  PP | 3230 (1110) |
  SP: 4 mg: number analyzed (Participants) | 0 | 1
  SP: 4 mg |  | 2170
  SP: 6 mg: number analyzed (Participants) | 0 | 5
  SP: 6 mg |  | 1600 (765)
  SP: 12 mg: number analyzed (Participants) | 0 | 3
  SP: 12 mg |  | 1840 (415)
  SP: 15 mg: number analyzed (Participants) | 0 | 3
  SP: 15 mg |  | 2150 (275)

18. Secondary Outcome: PAP: SP: Percent Change From Baseline in the 9-HPT to Week 104
Description: 9-HPT is a test of upper extremity (arm and hand) function.Participant is seated at table with small, shallow container holding pegs & block containing 9 empty holes.On start command (stopwatch started),participant picks up 9 pegs one at a time as quickly as possible, puts them in 9 holes & once they are in holes, removes them again as quickly as possible one at a time,replacing them into shallow container,2 consecutive trials of dominant hand followed immediately by 2 consecutive trials of non-dominant hand.Total time (ranging up to 300 seconds):averaged, converted to reciprocals which were averaged and back-transformed to obtain global 9-HPT.Higher value indicates higher disability.Baseline: last available value before or equal to first dose of study drug date in PAP.Secondary efficacy population:all enrolled participants with diagnosis of juvenile/adolescent late-onset GM2 gangliosidosis,GM1 gangliosidosis,saposin C deficiency,sialidosis type 1 or juvenile/adult galactosialidosis.
Time Frame: Baseline (Day 1) and Week 104
Population: as for outcome 10
Measure: Mean (Standard Error); unit: percent change
Arm/Group | PAP: SP: Venglustat
Number analyzed (Participants) | 11
percent change
  Juvenile/adolescent late-onset GM2 gangliodosis: number analyzed (Participants) | 4
  Juvenile/adolescent late-onset GM2 gangliodosis | -1.2 (24.5)
  GM1 gangliosidosis: number analyzed (Participants) | 6
  GM1 gangliosidosis | 11.7 (34.9)
  Sialidosis type 1: number analyzed (Participants) | 1
  Sialidosis type 1 | NA — Due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality.
  Juvenile/adult galactosialidosis: number analyzed (Participants) | 0
  Saposin C deficiency: number analyzed (Participants) | 0

19. Secondary Outcome: PAP: SP: Number of Participants With >=80% Compliance as Per Method of Intake
Description: For the secondary pediatric population, the acceptability and palatability of venglustat tablets was assessed through the route of venglustat administration collected in the electronic case report form and study drug compliance throughout PAP. The assessment was based on tablet always swallowed as whole or chewed and swallowed at least once. Number of participants with >=80% compliance for each is presented here.
Time Frame: Baseline (Day 1) to Week 104
Population: Secondary safety population included all enrolled participants with a clinical diagnosis of juvenile/adolescent late-onset GM2 gangliosidosis, GM1 gangliosidosis, saposin C deficiency, sialidosis type 1, or juvenile/adult galactosialidosis, who received at least 1 dose of study drug. Only pediatric participants were evaluated for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | PAP: SP: Venglustat
Number analyzed (Participants) | 13
Participants
  Participants always swallowed the tablet as whole: number analyzed (Participants) | 8
  Participants always swallowed the tablet as whole | 8
  Participants chewed and swallowed the tablet at least once: number analyzed (Participants) | 5
  Participants chewed and swallowed the tablet at least once | 4

ADVERSE EVENTS:
Time Frame: Adverse events:From first dose of study drug (Day 1) up to 104 weeks (PAP) and from 104 weeks up to 6 weeks post last drug in OLE, maximum duration 200 weeks due to study termination. Deaths were collected from first dose of study drug (Day 1) up to end of follow-up, maximum 200 weeks due to study termination.
Description: Analysis was performed on safety population (PAP: All enrolled participants who received at least 1 dose of study drug and OLE: all enrolled participants who received at least 1 venglustat dose after the 104-week visit).
Arm/Group | PAP: PP: Placebo | PAP: PP: Venglustat | PAP: SP: Venglustat | OLE: PP: Delayed Venglustat | OLE: PP: Early Venglustat | OLE: SP: Venglustat
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/40 | 1/16 | 1/16 | 0/34 | 0/14
Serious Adverse Events (participants affected / at risk) | 4/19 | 8/40 | 6/16 | 4/16 | 2/34 | 2/14
Other Adverse Events (participants affected / at risk) | 19/19 | 38/40 | 14/16 | 11/16 | 19/34 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAP: PP: Placebo (N=19) | PAP: PP: Venglustat (N=40) | PAP: SP: Venglustat (N=16) | OLE: PP: Delayed Venglustat (N=16) | OLE: PP: Early Venglustat (N=34) | OLE: SP: Venglustat (N=14)
Burn Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected Bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Completed Suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Persecutory Delusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal Achalasia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Mass (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAP: PP: Placebo (N=19) | PAP: PP: Venglustat (N=40) | PAP: SP: Venglustat (N=16) | OLE: PP: Delayed Venglustat (N=16) | OLE: PP: Early Venglustat (N=34) | OLE: SP: Venglustat (N=14)
Bacterial Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial Vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 3 (4) | 13 (14) | 7 (8) | 2 (2) | 2 (2) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (7)
Fungal Foot Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Helicobacter Gastritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected Bite (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Kidney Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (2) | 5 (13) | 2 (2) | 1 (3) | 1 (2)
Oral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Perichondritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (2) | 6 (9) | 2 (2) | 0 (0) | 3 (4) | 2 (2)
Urinary Tract Infection Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Iron Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (9) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Emotional Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Grief Reaction (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance Disorder (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Disturbance In Attention (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 10 (19) | 4 (10) | 2 (2) | 3 (3) | 1 (9)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyporeflexia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myasthenia Gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Speech Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cataract Cortical (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract Nuclear (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract Subcapsular (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid Ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lenticular Opacities (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meibomianitis (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual Field Defect (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Obstructive Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Colitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (6) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (8) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Duodenogastric Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastritis Erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 7 (10) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Tongue Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (5) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 7 (8) | 2 (3) | 3 (3) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Crystalluria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cervical Polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gait Disturbance (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Medical Device Site Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 3 (4) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Vaccination Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood Urine Present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression Rating Scale Score Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram Qt Prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte Count Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Strength Abnormal (Investigations) | 1 (8) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White Blood Cell Count Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 4 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (6) | 9 (10) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Face Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 10 (31) | 22 (61) | 2 (2) | 2 (3) | 4 (4) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immunisation Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was early terminated based on the absence of positive trends on clinical endpoints; there were no safety concerns. For sialidosis type 1 and juvenile/adult galactosialidosis, due to the rarity of the disease and the specificity of the endpoint, reporting individual-level data would risk compromising participant privacy and confidentiality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT04221451/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT04221451/SAP_001.pdf